CLINICAL TRIAL: NCT04386187
Title: Effects of the "Glutathione Support for Health (GSH)" Plan on Glutathione Status in Type 2 Diabetes
Brief Title: Glutathione-rich Foods for Type 2 Diabetes
Acronym: GSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ryan Bradley, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 180215
Record Dates: First submitted 2020-02-27; First posted 2020-05-13 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Glutathione; Nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a partial controlled-feeding trial in which participants will be initially randomized to a "food intervention" or "education control" and then will be crossed-over after 12 weeks.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Experimental Feeding (Experimental): Small glutathione-rich meals will be prepared and delivered to participants for 12 weeks.
  Interventions: Other: GSH Foods; Other: Nutrition education about glutathione sources in the diet
- Arm 2: Education Control (Active Comparator): Standard of care medical nutrition education for type 2 diabetes will be provided in the form of electronic handouts and web-based resources.
  Interventions: Other: Standard of care nutrition education for type 2 diabetes

INTERVENTIONS:
Other: GSH Foods — The intervention consists of customized foods/small meals that have been designed to be high in a single nutrient called glutathione (GSH).
  Arms: Arm 1: Experimental Feeding
Other: Nutrition education about glutathione sources in the diet — Four videos will outline food sources of glutathione, cooking methods to reduce systemic requirements for glutathione, food sources of nutrient cofactors for glutathione production and other related content.
  Arms: Arm 1: Experimental Feeding
Other: Standard of care nutrition education for type 2 diabetes — The educational control is provided with information on standard dietary interventions for diabetes as electronic handouts and web links.
  Arms: Arm 2: Education Control

SUMMARY:
The purpose of this research study is to find out whether certain plant-based foods may be beneficial for individuals with type 2 diabetes. To meet the goal, study participants will be fed known amounts of foods and nutrients. Before and after participants have eaten the food, they will self-measure height, weight, and waist circumference and study staff will administer questionnaires. Blood samples will be taken at a local lab to measure blood sugar and blood lipids.All study appointments will be conducted online.

DETAILED DESCRIPTION:
This research study is a randomized, controlled trial that will evaluate whether diet and nutrition education on, and short-term partial feeding of, specific plant foods high in the antioxidant glutathione will impact total glutathione status, gamma-glutamyltransferase (GGT) activity, glucose control or insulin sensitivity in people with type 2 diabetes. Dietary education will include information on plant sources of glutathione, as well as, cooking methods to reduce glycation and lipid peroxidation during cooking, which may indirectly alter glutathione status by reduce demand for elimination of these compounds. Participants will be randomized to one of two groups: the educational intervention plus partial feeding of two small meals per day vs. a wait list control group that will receive standard advice on nutrition for diabetes. After 12 weeks, the intervention group will no longer receive foods, but will be followed for 12 additional weeks to determine if lasting effects are achieved. After 12 weeks, the control group will receive access to the educational materials, but will not receive study foods, to see if the educational intervention alone impacts food/nutrition choices. Both groups will have lab measures (as described above) again after this additional 12 weeks, for a total duration of 24 weeks in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Ages 18 to 65
* Type 2 diabetes
* Free of self-reported acute and confounding chronic diseases (e.g., heart failure, kidney disease, liver disease, gastrointestinal disorder) based on a standardized medical history questionnaire
* Free of alcoholism, smoking and major cardiovascular event with the past 6 months
* Not on insulin to help manage diabetes
* Planning on staying in the San Diego area for the next 6 months
* Willing to select plant-based foods from a "menu" and eat the selected foods provided by the study team
* Have access to the internet and a computer
* Willing to view 4 weekly educational classes online, followed by periodic telephone and email contacts
* Agree to schedule and complete periodic questionnaires and measurements during up to four total online appointments

Exclusion Criteria:

* Alcoholism, smoking and recent cardiovascular events
* Individuals will be excluded if they report any dietary restrictions, allergies or preferences
* Unsuitability based on screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Total glutathione | 12 weeks
  Total glutathione concentration in the blood
gamma-glutamyltransferase (GGT) | 12 weeks
  Measure of glutathione demand in the blood

SECONDARY OUTCOMES:
Fasting glucose | 12 weeks
  Serum glucose concentration while fasting
Fasting insulin | 12 weeks
  Plasma insulin concentration while fasting
Hemoglobin A1c | 12 weeks
  Measure of glycemic control
Homeostasis Assessment Index of Insulin Resistance (HOMA-IR) | 12 weeks
  Estimate of insulin resistance
Low density lipoprotein concentration (LDL-c) | 12 weeks
  concentration of LDL lipoproteins in serum
High density lipoprotein concentration (HDL) | 12 weeks
  concentration of HDL lipoproteins in serum
Triglycerides | 12 weeks
  concentration of triglycerides in serum

OTHER OUTCOMES:
Total glutathione | 24 weeks
  Total glutathione concentration in the blood
gamma-glutamyltransferase (GGT) | 24 weeks
  Measure of glutathione demand in the blood
Fasting insulin | 24 weeks
  Plasma insulin concentration while fasting
Fasting glucose | 24 weeks
  Serum glucose concentration while fasting
Hemoglobin A1c | 24 weeks
  Measure of glycemic control
Homeostasis Assessment Index of Insulin Resistance (HOMA-IR) | 24 weeks
  Estimate of insulin resistance
Low density lipoprotein concentration (LDL-c) | 24 weeks
  concentration of LDL lipoproteins in serum
High density lipoprotein concentration (HDL) | 24 weeks
  concentration of HDL lipoproteins in serum
Triglycerides | 24 weeks
  concentration of triglycerides in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, ND, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No